CLINICAL TRIAL: NCT03161002
Title: Impact of Biomarkers on Pharmacokinetics and Pharmacodynamics of Ticagrelor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cui Yimin (Other)
Responsible Party: Sponsor-Investigator, Cui Yimin, Director of pharmacy，M.D & Ph.D, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Other Study IDs: 2016[1235]
Record Dates: First submitted 2017-05-09; First posted 2017-05-19 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Ticagrelor; Pharmacokinetics; Pharmacodynamics; Pharmacogenomics; Accurate Medication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- wild genotype: Through next generation sequencing, distinguish wild genotype of ticagrelor
  Interventions: Genetic: detection of genotype
- mutant genotype: Through next generation sequencing, distinguish mutant genotype of ticagrelor
  Interventions: Genetic: detection of genotype

INTERVENTIONS:
Genetic: detection of genotype — detection of genotype by next generation sequencing

SUMMARY:
It is general that there are many factors for individual differences of drugs in clinical application, of which genetic factors accounted for more than 20%. Ticagrelor is a new-type receptor antagonist of P2Y12 and it is not affected by the influence of CYP2C19 polymorphism. With lack of predicted biomarkers, especially the research data of Chinese, it has the important significance in studying individual differences of ticagrelor in the antiplatelet efficacy and safety, through the pharmacogenomics research.

The aim of this study is to determine the polymorphism of drug metabolizing enzymes, drug transporters and drug target genes in Chinese population. By detecting the gene polymorphism, we intend to study the pharmacokinetic/ pharmacodynamics/ pharmacogenomics (PK-PD-PG) correlation of ticagrelor and provide scientific basis for accurate medication guide for people to use ticagrelor.

ELIGIBILITY:
Inclusion Criteria:

(I)Chinese Healthy Volunteers

* In accordance with the inclusion criteria for each bioequivalence trial of ticagrelor;
* Sign informed consent of the research;
* Complete to collect indexes of pharmacodynamics and pharmacogenomics in the cycle with control drug.

(II)Chinese Patients

* With diagnosis of acute coronary syndrome (ACS), included unstable angina, non ST segment elevation myocardial infarction and ST segment elevation myocardial infarction;
* More than 18 years of age, male or female;
* Never received ticagrelor in a month and intend to take ticagrelor or have received ticagrelor for more than one week continuously；
* sign informed consent.

Exclusion Criteria:

(I)Chinese Healthy Volunteers

* In accordance with the exclusion criteria for each bioequivalence trial of ticagrelor;

(II)Chinese Patients

* With history of immunodeficiency disease, including positive HIV index;
* Positive Hepatitis B surface antigen (HBsAg) and HCV index;
* Combined therapy of CYP3A potent inhibitors (e.g., ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, Atazanavir, etc.), CYP3A substrate of narrow therapy window (e.g., cyclosporine, quinidine, etc.) and potent inducers of CYP3A (e.g., rifampin, phenytoin, carbamazepine, etc.) in 14 days before treatment with ticagrelor;
* Severe liver dysfunction and abnormal renal function;
* Uncontrolled hypertension, or systolic blood pressure > 180mmHg or diastolic pressure > 110mmHg during screening;
* Include contraindications of ticagrelor, such as hypersensitivity, active bleeding, moderate or severe liver disease, previous history of intracranial hemorrhage, gastrointestinal hemorrhage in the past 6 months and major operation within 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: (I)Chinese Healthy Volunteers：In accordance with the criteria of each bioequivalence trial of ticagrelor；150-200 cases (II)Chinese Patients：With diagnosis of acute coronary syndrome (ACS)，never received ticagrelor in a month and intend to take ticagrelor or have received ticagrelor for more than one week continuously；200 cases
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-05-31 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiac events (MACE) | At 1 year
  During the observation time, record the incidence of MACE after ticagrelor administration by telephone or outpatient clinic , including myocardial infarction, cardiac death, stent stenosis, stent thrombosis, ect.
Incidence of bleeding events | At 1 year
  During the observation time, record the incidence of bleeding events after ticagrelor administration by telephone or outpatient clinic, including subcutaneous bleeding, gingival bleeding, gastrointestinal bleeding, intracranial hemorrhage, etc.

SECONDARY OUTCOMES:
genotype detected by next generation sequencing | pre-dose of Ticagrelor
  Collect blood specimen before ticagrelor administration, then detect genotype of Ticagrelor by next generation sequencing.
Level of platelet reactivity assessed by ADP aggregation rate | At baseline, at 12 hours for Chinese healthy volunteers or at 48 hours for Chinese patients.
  Before and after ticagrelor administration, record the ADP aggregation rate detected by Light Transmittance Aggregometry(LTA).
Level of platelet reactivity assessed by PRI | At baseline, at 12 hours for Chinese healthy volunteers or at 48 hours for Chinese patients.
  Before and after ticagrelor administration, record PRI detected by VerifyNow System.
Expression level of miRNA | At baseline, at 12 hours for Chinese healthy volunteers or at 48 hours for Chinese patients.
  Before and after ticagrelor administration, detect the expression level of miRNA about pharmacodynamics.
Expression level of proteomics | At baseline, at 12 hours for Chinese healthy volunteers or at 48 hours for Chinese patients
  Before and after ticagrelor administration, detect the expression level of proteomics about pharmacodynamics
Expression level of LncRNA | At baseline, at 12 hours for Chinese healthy volunteers；at 48 hours for Chinese patients.
  Before and after ticagrelor administration, detect the expression level of LncRNA about pharmacodynamics.
Incidence of MACEs in the other observation times | At 1 month, 6 months and 2 years (according the actual duration of ticagrelor taken in patiens)
  During the other observation time, record the incidence of MACE after ticagrelor administration by telephone or outpatient clinic , including myocardial infarction, cardiac death, stent stenosis, stent thrombosis, ect.
Incidence of bleeding events in the other observation times | At 1 month, 6 months and 2 years (according the actual duration of ticagrelor taken in patiens)
  During the other observation time, record the incidence of bleeding events after ticagrelor administration by telephone or outpatient clinic, including subcutaneous bleeding, gingival bleeding, gastrointestinal bleeding, intracranial hemorrhage, etc.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Anhui Provincial Hospital（The First Affiliated Hospital Of USTC）, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - 900 Hospital of the Joint Logistics Team (Original name: Fuzhou General Hospital of Nanjing Militray Command), Fuzhou, Fujian
  - The 7th People's Hospital Of Zhengzhou, Zhengzhou, Henan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi

REFERENCES:
- [Derived] Xiang Q, Liu Z, Mu G, Xie Q, Zhang H, Zhou S, Wang Z, Guo N, Huang J, Jiang J, Li J, Yang G, Cui Y. Effect of Genetic Polymorphism Including NUP153 and SVEP1 on the Pharmacokinetics and Pharmacodynamics of Ticagrelor in Healthy Chinese Subjects. Clin Drug Investig. 2022 May;42(5):447-458. doi: 10.1007/s40261-022-01154-6. Epub 2022 Apr 30. PMID 35501592
- [Derived] Yuan D, Shi X, Gao L, Wan G, Zhang H, Yang Y, Zhao Y, Sun D. Identification of Potential Biological Factors Affecting the Treatment of Ticagrelor After Percutaneous Coronary Intervention in the Chinese Population. Pharmgenomics Pers Med. 2022 Jan 20;15:29-43. doi: 10.2147/PGPM.S338287. eCollection 2022. PMID 35082514